CLINICAL TRIAL: NCT06124664
Title: Study of Venous Outflow From the Lower Limbs in Patients With Pelvic Varicosities as a New Strategy for Compression Treatment of Pelvic Varicose Veins and Varicose Veins of the Lower Limb
Brief Title: Study of Venous Outflow From the Lower Limbs in Patients With Pelvic Varicosities
Status: Recruiting | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Sergey Gavrilov, MD, PhD, Clinical Professor, Pirogov Russian National Research Medical University
Other Study IDs: 012012548112
Record Dates: First submitted 2023-10-29; First posted 2023-11-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Varices; Varicose Veins of Lower Limb; Pelvic Pain Syndrome; Pelvic Congestive Syndrome
Keywords: pelvic varicose vein; venous outflow; chronic venous disease; compression treatment; duplex ultrasound; single-photon emission computed tomography
MeSH Terms: interventions — Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic pelvic varicose veins (PVV): 40 patients will include patients with symptomatic PVV (pelvic pain, dyspareunia, heaviness in the hypogastrium) and without symptoms and signs of CVD.
  Interventions: Diagnostic Test: Radionuclide venography; Diagnostic Test: single-photon emission computed tomography
- Asymptomatic PVV: 40 pdtients will consist of women with asymptomatic PVV with signs of CVD.
  Interventions: Diagnostic Test: Radionuclide venography; Diagnostic Test: single-photon emission computed tomography
- varicose veins of the lower limb: 10 patients with varicose veins of the lower limb without PVV and pelvic congestion syndrome (PCS)
  Interventions: Diagnostic Test: Radionuclide venography; Diagnostic Test: single-photon emission computed tomography

INTERVENTIONS:
Diagnostic Test: Radionuclide venography — With the patient in an upright position, 370 MBq of 99mTc pertechnetate is injected into one of the dorsal veins of the foot after applying a tourniquet in the area of the ankle joint. Then, with the help of a gamma camera detector, the movement of the radiopharmaceutical is monitored in the following segments: tibial (muscular-venous pump of the lower leg), popliteal, femoral and iliocaval. To study the evacuation function of the muscular-venous pump (MVP) of the leg, using an analytical computer program, areas of interest are identified in the tendon, muscle parts of the veins of the leg and the popliteal vein. The time of evacuation of the radiopharmaceutical from the MVP of the leg is estimated - the average transport time of the isotope.
Diagnostic Test: single-photon emission computed tomography — SPECT of the pelvic veins with in vivo-labelled red blood cells (RBCs). For radionuclide assessment of the state of the pelvic veins, 2 ml of Perfotech solution is injected into the cubital vein for subsequent "labeling" of red blood cells in vivo. In 20 minutes. 370 MBq of 99mTc-pertechnetate is injected into one of the veins of the dorsum of the foot and radionuclide venoscintigraphy is performed according to the method presented above. 20 minutes after the administration of the radiopharmaceutical and the venography, SPECT of the pelvic veins is performed. Tomography of the distribution of labeled erythrocytes in the pelvic veins is carried out in a circular orbit with the gamma camera detector rotated 360°. The analysis of the obtained information is carried out using the standard ECT Protocol software package, which allows obtaining sections in 3 projections (sagittal, transversal and coronal) with a slice step of 8 mm.

SUMMARY:
Compression therapy is basic treatment for chronic venous disease (CVD) of the lower limbs. Numerous studies have demonstrated the efficacy and safety of compression therapy in relieving symptoms such as pain, venous edema, leg heaviness and fatigue, as well as accelerating the healing of venous ulcers. It has been established that сompression therapy is indicated for patients with both minimally expressed manifestations of CVD and severe forms of the disease. At the same only one study has been conducted to assess the correction of venous outflow from the lower limbs and pelvis in patients with pelvic varicose vein (PVV) and pelvic congestion syndrome (PCS). However, the incidence of this pathology ranges from 15 to 30% in the female population. The cost to the healthcare system of treating these patients in the United States exceeds $2 billion. To date, the options and indications for compression therapy in patients with concomitant PVV and CVD have not been defined. The rational use of compression in this cohort of patients may contribute to the improvement of effective conservative treatment. In addition, inappropriate prescription of compression to patients with pelvic venous disease (which can be observed in real clinical practice) may discredit this simple, effective and safe therapeutic method. In addition, the research devoted to the problem of compression treatment of PVV will contribute to the development of new special compression products aimed at accelerating venous outflow from the pelvic organs. It can be assumed that this will serve as a stimulus for obtaining new data on the therapeutic effects of compression and create conditions for the creation of new technological directions in the production of compression knitwear.

DETAILED DESCRIPTION:
This is a single-center, prospective, comparative cohort study. The duration of the study is from 4/5/2023 to 1/12/2023. The study will include 90 patients (40 patients with symptomatic PVV without CVD, 40 patients with asymptomatic PVV and symptoms of CVD, 10 patients with CVD of the lower limb without PVV.

Currently, the term "varicose veins" implies not only the pathology of the superficial veins of the lower limbs, but also the pelvic veins. As yet, no epidemiological studies have investigated the frequency of the combination of pelvic and lower limb varicose veins, but in some studies the authors point to a combination of lower limb varicose veins and pelvic varicose veins (PVV) in 30-60% of patients. In this scenario, we are discussing the disease's clinically manifested forms, where lower limb varicose veins are visually identified and pelvic veins are identified by ultrasound and manifest as symptoms of pelvic congestion syndrome. There is no evidence of a concomitant occurrence of asymptomatic or latent forms of varicose veins in the lower limbs and PVV. (In this cases during duplex ultrasound angioscanning (DUS), pathological blood reflux is detected in the dilated superficial veins of the lower limbs and pelvis. However, there are no symptoms or signs of the disease.) As a result, it is not possible to assess the true prevalence of the combination of CVD and PVV.

At the same time, it is evident that dilatation and reflux in pelvic veins cannot but affect the clinical course of CVD in general and lower limb varicose vein disease in particular. Multiple studies from our clinic and foreign colleagues have substantiated this claim. It is caused not only by anatomical links between pelvic veins and lower limbs (perineal, clitoral perforating veins, tributaries of internal iliac veins), but also by common triggering mechanisms and similar pathogenesis of lower limb varicose vein disease and PVV.

Considering the above, valid questions arise about the effect of pelvic varicose veins with reflux on lower extremity venous outflow:

1. How does asymptomatic pelvic vein dilation with reflux impact venous outflow from the lower extremities and the clinical manifestations of CVD?
2. Does symptomatic pelvic vein dilation with reflux affect venous outflow from the lower limbs and clinical manifestations of CVD?
3. Does vulvar vein dilation affect venous outflow from the lower limbs and CVD clinical manifestations?
4. Is the severity or exposure of pelvic congestion syndrome a predictor for the development of lower limb venous outflow disorders?
5. How does the severity of clinical manifestations of PCS correspond to the severity of hemodynamic disturbance, as determined through instrumental research methods?

These questions have significance not only in academic and scientific domains. They are directly related to the strategy and tactics of treating patients with a combination of varicose veins of lower limbs and PVV, PCS and CVD, since the following fundamental issues have not yet been resolved:

1. Do asymptomatic patients with instrumental detection of PVV and lower limb varicose vein require correction?
2. Is it appropriate to utilize compression knitwear in patients with an asymptomatic course of instrumentally confirmed venous outflow disorders with a combination of pelvic and lower extremity varicose veins?
3. Can the coefficient of pelvic venous congestion be utilized as a quantitative indicator to prescribe compression treatment for venous outflow disorders in the lower limbs of asymptomatic patients without signs of CVD? In other words, can the coefficient of pelvic venous congestion be used as a reference index for correcting the evacuative function of the tibial MVP in patients without clinical manifestations of CVD?
4. How effective is compression in correcting impaired venous outflow from the lower limbs in PVV patients? The severity of the clinical course of lower limb CPV is determined by objective symptoms such as pain, edema, trophic disorders, and venous ulceration. In patients with CVD, the severity of the disease course determines the development of pelvic congestion syndrome (PCS), which is manifested by chronic pelvic pain (CPP), hypogastric heaviness, and dyspareunia. CPP and dyspareunia are the main indicators of the severity of the clinical course of PCS. It has been demonstrated that PCS exacerbates the symptoms of CVD. Thus, correlating the severity of pelvic pain to the degree of pelvic venous fullness (coefficient calculated by pelvic venous scintigraphy) allows us to assume the presence of venous outflow disorders of the lower extremities. According to this hypothesis, the presence and severity of venous outflow disorders of the lower limbs can be determined not only by the results of instrumental examination of the pelvic and limb veins, but also by clinical assessment of the severity of CPP.

ELIGIBILITY:
Inclusion Criteria:

* Patient age from 18 to 40 years;
* Presence of pelvic varicose veins according to DUS data;
* Reflux in the pelvic veins for more than 1 second before this DUS;
* Reflux in the superficial veins of the lower limbs.

Exclusion Criteria:

* Menopause;
* Pregnancy;
* Postthrombotic disease;
* Suspicion of May-Turner syndrome;
* Ultrasound signs of nutcracker syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patient age from 18 to 40 years and who regardless of their sex assigned at birth, identifies as a woman.
Study Population: The study will consecutively include 90 female patients, including 80 patients with PVV and 10 patients without PVV. All patients will have a clinical examination and DUS of the veins of the pelvis and lower limbs, regardless of the presence or absence of clinical manifestations of diseases of the veins of the pelvis and lower limbs. Аll patients were performed radionuclide venography of the lower limbs and emission computed tomography (SPECT) of the pelvic veins with in vivo-labelled red blood cells (RBCs). Based on the results of radionuclide venography and SPECT, quantitative indicators of the work of the lower limbs MVP will be calculated (average transport time RPH) and Cpvc.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
The average transport time of the isotope | Day 0 and Day 10
  Average transport time of the isotope is a value inversely proportional to the volumetric velocity of blood flow. The greater the average transport time of the isotope, the slower the speed of blood flow through the deep veins of the leg and vice versa. In addition, the linear speed of blood flow through the tibial veins is calculated. The data obtained allow us to judge the function of the MVP of the lower leg.
coefficient of the pelvic venous congestion | Day 0
  The computer equipment of the gamma camera allows you to calculate the number of pulses from the area of interest. The radiopharmaceutical radiation activity is recorded by the gamma camera in pulses per second. Pulse per second is a quantitative expression of the content of labeled red blood cells in the area of interest. Taking into account the different speed of blood flow in the pelvic veins in different patients and in order to objectify the data obtained, the ratio of pulse counts from 2 standard areas of interest is used - the veins of the uterus and parametrium and the common iliac vein on either side. This ratio is called coefficient of the pelvic venous congestion(Сpvc). The activity of labeled erythrocytes in this vessel is the most stable value. The activity of erythrocyte-phosphate-pertechnetate complexes in the venous plexuses depends on the presence of their varicose transformation and the deposition of blood in them.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia V Koroleva, PhD, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Ananstsia Grishenkova, Moskva, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Partsch H. Compression for the management of venous leg ulcers: which material do we have? Phlebology. 2014 May;29(1 suppl):140-145. doi: 10.1177/0268355514528129. Epub 2014 May 19. PMID 24843100
- [Result] Vin F, Benigni JP; International Union of Phlebology; Bureau de Normalisation des Industries Textiles et de l'Habillement; Agence Nationale d'Accreditation et d'Evaluation en Sante. Compression therapy. International Consensus Document Guidelines according to scientific evidence. Int Angiol. 2004 Dec;23(4):317-45. No abstract available. PMID 15767979
- [Result] Nicolaides A, Kakkos S, Eklof B, Perrin M, Nelzen O, Neglen P, Partsch H, Rybak Z. Management of chronic venous disorders of the lower limbs - guidelines according to scientific evidence. Int Angiol. 2014 Apr;33(2):87-208. No abstract available. PMID 24780922
- [Result] Gavrilov SG, Karalkin AV, Turischeva OO. Compression treatment of pelvic congestion syndrome. Phlebology. 2018 Jul;33(6):418-424. doi: 10.1177/0268355517717424. Epub 2017 Jun 22. PMID 28639874
- [Result] Gultasli NZ, Kurt A, Ipek A, Gumus M, Yazicioglu KR, Dilmen G, Tas I. The relation between pelvic varicose veins, chronic pelvic pain and lower extremity venous insufficiency in women. Diagn Interv Radiol. 2006 Mar;12(1):34-8. PMID 16538582
- [Result] Whiteley AM, Taylor DC, Dos Santos SJ, Whiteley MS. Pelvic venous reflux is a major contributory cause of recurrent varicose veins in more than a quarter of women. J Vasc Surg Venous Lymphat Disord. 2014 Oct;2(4):411-5. doi: 10.1016/j.jvsv.2014.05.005. Epub 2014 Jun 24. PMID 26993547
- [Result] Bora A, Avcu S, Arslan H, Adali E, Bulut MD. The relation between pelvic varicose veins and lower extremity venous insufficiency in women with chronic pelvic pain. JBR-BTR. 2012 Jul-Aug;95(4):215-21. doi: 10.5334/jbr-btr.623. PMID 23019985

DOCUMENTS (1):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT06124664/Prot_000.pdf